CLINICAL TRIAL: NCT05975320
Title: "ORBIT" Versus "HAS-BLED" Scores in Predicting Major Bleeding in Patients With Atrial Fibrillation Receiving Oral Anticoagulants.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Yasmin Mohamed Mohamed, resident of internal medicine department, Sohag university hospital, Sohag University
Other Study IDs: Soh-med-23-07-03MS
Record Dates: First submitted 2023-07-27; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Patients With Atrial Fibrillation Receiving Oral Anticoagulants
MeSH Terms: interventions — Warfarin; apixaban

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Warfarin — Patients receiving oral anticoagulants will be followed up for 6 months to detect occurrence of any major bleeding events include (spontaneous epistaxis , spontaneous bleeding per gums , hematemesis , bleeding per rectum , intracranial hemorrhage and internal hemorrhage ). Then, incidence of bleeding events using both (HAS-BLED) & (ORBIT) SCORES will be calculated and compared for all cases .
  Other Names: apixaban, Rivarospire

SUMMARY:
Atrial fibrillation (AF) is type of arrhythmia characterized by an irregular and often rapid heartbeats, it has strong associations with other cardiovascular diseases, such as heart failure, coronary artery disease (CAD), valvular heart disease, diabetes mellitus, thyrotoxicosis and hypertension.

Atrial fibrillation is the most frequent cardiac arrhythmia. It has been estimated that 6-12 million people worldwide will suffer this condition in the US by 2050 and 17.9 million people in Europe by 2060. Atrial fibrillation is a major risk factor for ischemic stroke and provokes important economic burden along with significant morbidity and mortality .

(AF) is arrhythmia with the potential to cause thromboembolism. Studies suggest that AF increases the risk of stroke five-folds. Stroke prevention is central to the management of patients with atrial fibrillation (AF), and effective stroke prevention requires oral anticoagulation (OAC). Either a vitamin K antagonist (VKA; e.g. warfarin) or a non-VKA oral anticoagulant (NOAC) .

It's essential reach the balance between prevention of thromboembolic as well as bleeding events during the anticoagulant use.

ELIGIBILITY:
Inclusion Criteria:

* All patients with atrial fibrillation :

  1. Aged 18 years old or older .
  2. Underwent cardiac valve replacement
  3. Who have valvular heart disease receiving anticoagulants .
  4. Who have non valvular AF in whom CHA2DS 2VASc score 2 or more.
  5. Receiving either vitamin K antagonist e.g warfarin or NOAC .

Exclusion Criteria:

1. Patients age less than 18 years old
2. Patients receiving anticoagulants without atrial fibrillations
3. Pregnant patients with AF
4. Patients with AF on Non oral anticoagulants

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: -All patients with atrial fibrillation :
  1. Aged 18 years old or older .
  2. Underwent cardiac valve replacement
  3. Who have valvular heart disease receiving anticoagulants .
  4. Who have non valvular AF in whom CHA2DS 2VASc score 2 or more.
  5. Receiving either vitamin K antagonist e.g warfarin or NOAC .
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
incidence of bleeding events using both (HAS-BLED) & (ORBIT) SCORES | 6 months
  Patients receiving oral anticoagulants will be followed up for 6 months to detect occurrence of any major bleeding events include (spontaneous epistaxis , spontaneous bleeding per gums , hematemesis , bleeding per rectum , intracranial hemorrhage and internal hemorrhage ). Then, incidence of bleeding events using both (HAS-BLED) & (ORBIT) SCORES will be calculated and compared for all cases .

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Piccini JP, Fraulo ES, Ansell JE, Fonarow GC, Gersh BJ, Go AS, Hylek EM, Kowey PR, Mahaffey KW, Thomas LE, Kong MH, Lopes RD, Mills RM, Peterson ED. Outcomes registry for better informed treatment of atrial fibrillation: rationale and design of ORBIT-AF. Am Heart J. 2011 Oct;162(4):606-612.e1. doi: 10.1016/j.ahj.2011.07.001. PMID 21982650
- [Background] Pisters R, Lane DA, Nieuwlaat R, de Vos CB, Crijns HJ, Lip GY. A novel user-friendly score (HAS-BLED) to assess 1-year risk of major bleeding in patients with atrial fibrillation: the Euro Heart Survey. Chest. 2010 Nov;138(5):1093-100. doi: 10.1378/chest.10-0134. Epub 2010 Mar 18. PMID 20299623
- [Background] De Caterina R, Husted S, Wallentin L, Andreotti F, Arnesen H, Bachmann F, Baigent C, Huber K, Jespersen J, Kristensen SD, Lip GY, Morais J, Rasmussen LH, Siegbahn A, Verheugt FW, Weitz JI. Vitamin K antagonists in heart disease: current status and perspectives (Section III). Position paper of the ESC Working Group on Thrombosis--Task Force on Anticoagulants in Heart Disease. Thromb Haemost. 2013 Dec;110(6):1087-107. doi: 10.1160/TH13-06-0443. Epub 2013 Nov 14. PMID 24226379
- [Background] O'Brien EC, Simon DN, Thomas LE, Hylek EM, Gersh BJ, Ansell JE, Kowey PR, Mahaffey KW, Chang P, Fonarow GC, Pencina MJ, Piccini JP, Peterson ED. The ORBIT bleeding score: a simple bedside score to assess bleeding risk in atrial fibrillation. Eur Heart J. 2015 Dec 7;36(46):3258-64. doi: 10.1093/eurheartj/ehv476. Epub 2015 Sep 29. PMID 26424865